CLINICAL TRIAL: NCT07041957
Title: Biphasic Positive Airway Pressure Ventilation Versus Flow-Controlled Ventilation in Burn Patients: A Monocentric, Randomized Controlled, Parallel Group Trial
Brief Title: Biphasic Positive Airway Pressure Ventilation Versus Flow-Controlled Ventilation in Burn Patients
Acronym: BIFLOWBURN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bergmannsheil Bochum (Other)
Collaborators: Department of Plastic, Reconstructive and Burn Surgery, BG University Hospital Bergmannsheil, Ruhr University Bochum, Bochum, Germany (Unknown); Department of Medical Informatics, Biometry and Epidemiology, Ruhr University Bochum, Bochum, Germany (Unknown); Medical Proteom-Center (MPC), Ruhr University Bochum, Bochum, Germany (Unknown); Department of Anesthesiology, Intensive Care and Pain Medicine, BG University Hospital Bergmannsheil, Ruhr University Bochum (Unknown); Department of Anesthesiology, Intensive Care, Pain and Palliative Care, Marien Hospital Herne, Ruhr University Bochum, Bochum, Germany (Unknown)
Responsible Party: Principal Investigator, Simon Becker, Jun.-Prof. Dr. med. Simon Becker, M.D., University Hospital Bergmannsheil Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-7944; 23-7944 (Other Grant/Funding Number: Department of Anesthesiology and Intensive Care Medicine, University Hospital Bergmannsheil, Ruhr University Bochum)
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Burn Injury; Inhalational Injury; Pulmonary Complications; Ventilator-induced Lung Injury (VILI)
Keywords: Flow-controlled ventilation; Pressure-controlled ventilation; Mechanical Power; Dissipated Energy; Ventilator-induced lung injury
MeSH Terms: conditions — Burns; Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to different ventilators during the interventions, outcome assessors can only be blinded after intervention withdrawal. Participants are blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flow-Controlled Ventilation (Experimental): Individualized flow-controlled ventilation (FCV) with a compliance-guided positive end-expiratory pressure (PEEP), a compliance-guided driving pressure (ΔP) resulting in a liberal tidal volume, and adjustment of airway flows and respiratory rates being required for normocapnia.
  Interventions: Other: Individualized flow-controlled ventilation strategy
- Pressure-Controlled Ventilation via Biphasic Positive Airway Pressure Ventilation (Active Comparator): Conventional pressure-controlled ventilation via application of Biphasic Positive Airway Pressure (BIPAP) ventilation with a compliance-guided positive end-expiratory pressure (PEEP), a driving pressure (ΔP) for a tidal volume of 6-8 ml/kg predicted body weight, and adjustment of respiratory rates being required for normocapnia but no adjustment/control of airway flows.
  Interventions: Other: Pressure-controlled ventilation strategy via the application of Biphasic Positive Airway Pressure ventilation

INTERVENTIONS:
Other: Individualized flow-controlled ventilation strategy — 1. Compliance-guided PEEP trial: An incremental PEEP trial from 5 to 15 cmH2O in 2 cmH2O steps with a constant driving pressure (ΔP) will be performed. At the first PEEP level, the tidal volume is set to 6-8 ml/kg PBW. The best PEEP level is defined as the one with the highest dynamic compliance. Participants are ventilated with this PEEP level + 1-2 cmH2O for a reduction of lung de-recruitment and atelectrauma.
  2. Compliance-guided driving pressure (ΔP) trial: In the FCV group, an additional incremental ΔP trial in 1 cmH2O steps is initiated after the PEEP trial. This trial evaluates if the tidal volume increases (over-)proportional to the dynamic compliance on the previous ΔP level when the ΔP is increased by 1 cmH2O. In the FCV group, participants are ventilated with a ΔP consistent with the highest dynamic compliance ± 1-2 cmH2O. The compliance-guided PEEP and ΔP trials are repeated every 8 hours in order to account for changes in overall lung compliance.
  Other Names: FCV
  Arms: Flow-Controlled Ventilation
Other: Pressure-controlled ventilation strategy via the application of Biphasic Positive Airway Pressure ventilation — 1. Compliance-guided PEEP trial: An incremental PEEP trial from 5 to 15 cmH2O in 2 cmH2O steps with a constant driving pressure (ΔP)will be performed. At the first PEEP level, the tidal volume is set to 6-8 ml/kg PBW. The best PEEP level is defined as the one with the highest dynamic compliance. Participants are ventilated with this PEEP level + 1-2 cmH2O for a reduction of lung de-recruitment and atelectrauma.
  2. The driving pressure (ΔP) is set to achieve a tidal volume of 6-8 ml/kg predicted body weight.
  The compliance-guided PEEP trial is repeated every 8 hours in order to account for changes in overall lung compliance.
  Other Names: PCV via BIPAP
  Arms: Pressure-Controlled Ventilation via Biphasic Positive Airway Pressure Ventilation

SUMMARY:
The goal of this clinical trial is to learn if the new ventilation mode flow-controlled ventilation (FCV) is a more protective mode of ventilation for adult patients after severe burn injury. The main question it aims to answer is:

Does FCV reduce the mechanical power (a key determinant of ventilator-induced lung injury) compared to conventional pressure-controlled ventilation (PCV) during ventilation of patients with burn injury?

Researchers will compare FCV with PCV for up to 70 hours of ventilation to see if the mechanical power is reduced during ventilation of participants being in need of ventilation after severe burn injury.

Ventilation of participants will be controlled by either FCV or PCV. Group-specific ventilation will have the following characteristics:

* FCV: Control of airway flows during inspiration and expiration, use of individualized lower and upper airway pressures and no fixed values for the volumes being inspired and expired (tidal volumes)
* PCV: No control of airway flows during expiration, use of individualized lower airway pressures and upper airway pressures for a fixed tidal volume during each breath (6-8 ml/kg ideal body weight)

In total, at least 24 participants in need of ventilation after severe burn injury will be ventilated either with FCV (12 participants) or PCV (12 participants) for up to 70 hours.

During ventilation mechanical power is computed according to certain ventilation parameters. Additionally, we evaluate organ functions of the cardiovascular systems, the lungs and other organs during and after the group-specific ventilation.

DETAILED DESCRIPTION:
Invasive ventilation can cause ventilator-induced lung injury. There is growing evidence that high mechanical power during (prolonged) controlled ventilation is associated with ventilator-induced lung injury and pulmonary complications.

Large animal model and perioperative clinical trial data have shown that the individualized application of the flow-controlled ventilation (FCV) mode can reduce mechanical power compared to conventional pressure-controlled ventilation (PCV).

Burn patients with or without inhalational injury are at high risk of pulmonary complications like pneumonias or the acute respiratory distress syndrome due to the hyperinflammatory state and also the intensive care treatment after a burn injury. If these patients need mechanical ventilation, this might aggravate lung injury.

With the study BIFLOWBURN we want to test the hypothesis that the mechanical power during controlled ventilation of burn patients is reduced with the individualized application of FCV compared to conventional PCV via Biphasic Positive Airway Pressure (BIPAP) ventilation.

BIFLOWBURN is a single-center, randomized, parallel-group trial with two intervention arms:

* Controlled BIPAP ventilation (n=12) with a compliance-guided positive end-expiratory pressure (PEEP) and driving pressure (ΔP) for tidal volumes of 6-8 ml/kg predicted body weight compared to
* optimized FCV (n=12) with a compliance-guided PEEP and a compliance-guided ΔP, resulting in liberal tidal volumes.

The group-specific controlled ventilation mode will be applied for a maximum of 70 hours.

As the primary study endpoint, the mechanical power in joules per minute (J/min) is computed during group-specific controlled ventilation.

As secondary study aims, clinically relevant patient outcomes are analyzed as explorative secondary outcomes, e.g., lung function, ventilatory parameters, the incidences of pulmonary and extra-pulmonary complications as well as different intensive care scores for the assessment of organ dysfunctions.

As an additional sub-study with an exploratory approach, parameters of different advanced haemodynamic monitoring techniques are assessed. Within a further ancillary study, biomarkers of acute lung injury and/or the burn inhalational injury will be characterized by molecular biological methods.

BIFLOWBURN is the first randomized controlled trial which assesses mechanical power during the ventilation of burn patients by comparing the alternative mode of flow-controlled ventilation with a conventional ventilation mode.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg
* Invasive ventilation time ≤ 24 hours before admission to the burn ICU or indication for intubation and invasive ventilation within 48 hours after admission to the burn ICU
* Estimated (further) invasive ventilation time ≥ 24 hours
* Intervention start within 48 hours after admission to the burn ICU
* Establishment of a central venous line and invasive blood pressure monitoring as part of the intensive care therapy before the intervention start
* Signed informed consent from the participant, legal guardian, next of kin in incompetent patients, or an intensivist in charge and independent from the Trial Management Committee in incompetent patients without a representative of the patients will

Exclusion Criteria:

* Participation in another interventional trial
* Duration of invasive ventilation > 24 hours at the time point of admission to the burn ICU
* Estimated (further) invasive ventilation time < 24 hours
* Patients being treated in the burn ICU for (suspected) severe skin reactions such as Stevens-Johnson syndrome (SJS) or toxic epidermal necrolysis (TEN)
* Lack of consent from the participant, legal guardian, next of kin, or intensivist in charge to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mechanical power | Mechanical power will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  We will compute mechanical power in joules per minute (J/min) hourly according to the surrogate formulae [Minute ventilation * (Peak airway pressure + PEEP + Inspiratory flow/6)]/20 for FCV and 0.098 * respiratory rate * tidal volume * [PEEP + ΔP] for PCV/BIPAP

SECONDARY OUTCOMES:
Dissipated energy/power | The dissipated energy/power will be assessed at least hourly/continously during up to 70 hours of controlled, group-specific ventilation.
  The hysteresis of the pressure-volume loop represents the dissipated energy in joules, that is dissipated during one ventilation cycle. The dissipated power per unit time can be computed by the respiratory rate per unit time, e.g. Joules per minute (J/min).
Respiratory rate | Respiratory rates will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Respiratory rate per minute
Tidal volume | Tidal volumes will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Tidal volume in ml
Minute volume | Minute volumes will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Minute volume in liter per minute
Airway pressures | Airway pressures will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Airway pressures like positive end-expiratory pressure (PEEP), peak airway pressure, driving pressure (ΔP) and mean airway pressure in cmH2O
Dynamic compliance | Dynamic compliances will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Dynamic compliance in ml per cmH2O will be calculated according to the formula tidal volume/driving pressure.
Airway resistance | Airway resistances will be assessed hourly during up to 70 hours of controlled, group-specific ventilation.
  Airway resistance in cmH2O/L/s as displayed on the ventilator.
Oxygenation indices | Oxygenation indices will be assessed every 4-8 hours with arterial blood gas analyses during up to 70 hours of controlled, group-specific ventilation.
  Computed as partial pressure of arterial oxygen/inspired oxygen fraction
Pulmonary complications | Pulmonary complications will be assessed within the first ten days after randomization.
  Incidence of pulmonary complications including but not limited to need for non-invasive ventilation / high flow nasal cannula therapy, reintubation, tracheotomy, prone positioning, ARDS, pleural effusions, pneumothorax, bronchoscopy, suspected or confirmed pneumonia
Extra-pulmonary complications | Extra-pulmonary complications will be assessed within the first ten days after randomization.
  Incidence of extra-pulmonary complications including but not limited to systemic inflammatory response syndrome (SIRS), sepsis, septic shock, new arrythmias, cardiac arrest, infection other than pneumonia treated with antibiotics, delirium, acute kidney injury
Sequential Organ Failure Assessment (SOFA) Score | The Sequential Organ Failure Assessment (SOFA) Score will be assessed daily within the first ten days after randomization.
  The Sequential Organ Failure Assessment (SOFA) Score ranges from zero (no organ failure present) to 24 (most severe failure in all assessed organ systems).
Lung Injury Score (Murray) | The Lung Injury Score will be assessed daily within the first ten days after randomization.
  The Murray Score for Acute Lung Injury is ranging from zero (no lung injury) to 16 (most severe lung injury).
Acute Physiology and Chronic Health Evaluation (APACHE) Score | The Acute Physiology and Chronic Health Evaluation (APACHE) Score will be assessed daily within the first ten days after randomization.
  The Acute Physiology and Chronic Health Evaluation (APACHE) Score provides an estimate of in-hospital ICU mortality with lower score values being associated with a lower mortality rate and higher score values being associated with a higher mortality rate.
Duration of invasive ventilation | Participants will be followed-up on length of invasive ventilation for 6 months after the interventions.
  The total length of invasive ventilation will be assessed in minutes.
Length of stay | Participants will be followed-up for 6 months after the interventions.
  Participant will be monitored on ICU and hospital length of stay in days.
Mortality | Participants will be followed-up for 6 months after the interventions.
  Mortality of participants will be monitored up to 6 months after the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Peter K. Zahn, Prof. Dr. med., M.D., Study Director — Ruhr University Bochum, BG University Hospital Bergmannsheil, Department of Anesthesiology, Intensive Care and Pain Medicine; Simon Becker, Jun.-Prof. Dr. med., M.D., Principal Investigator — Ruhr University Bochum, BG University Hospital Bergmannsheil, Department of Anesthesiology, Intensive Care and Pain Medicine
Locations (1):
- BG University Hospital Bergmannsheil, Ruhr University Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
Before the enrolment of the last participant, the study protocol including the statistical analysis plan will be published in an appropriate journal after peer-reviewing.
  After pseudonymisation, data is transferred and processed with the web-based application software REDCap™. This enables data sharing of complete deidentified data sets of all primary and secondary study outcome data with the scientific community upon personal request with a reasonable proposal to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning immediately after publication of the respective main study and explorative ancillary studies with no end date.
Access Criteria: IPD can be accessed by peers and other investigators upon personal request to the principal investigator with a reasonable proposal including a detailed description of the planned analyses. The Trial Management Committee will critically review this proposal together with the principal investigator.

REFERENCES:
- [Background] Bittner E, Sheridan R. Acute Respiratory Distress Syndrome, Mechanical Ventilation, and Inhalation Injury in Burn Patients. Surg Clin North Am. 2023 Jun;103(3):439-451. doi: 10.1016/j.suc.2023.01.006. Epub 2023 Mar 21. PMID 37149380
- [Background] Van Oosten JP, Francovich JE, Somhorst P, van der Zee P, Endeman H, Gommers DAMPJ, Jonkman AH. Flow-controlled ventilation decreases mechanical power in postoperative ICU patients. Intensive Care Med Exp. 2024 Mar 19;12(1):30. doi: 10.1186/s40635-024-00616-9. PMID 38502268
- [Background] Spraider P, Abram J, Martini J, Putzer G, Glodny B, Hell T, Barnes T, Enk D. Flow-controlled versus pressure-controlled ventilation in cardiac surgery with cardiopulmonary bypass - A single-center, prospective, randomized, controlled trial. J Clin Anesth. 2023 Dec;91:111279. doi: 10.1016/j.jclinane.2023.111279. Epub 2023 Oct 3. PMID 37797394
- [Background] Abram J, Martini J, Spraider P, Putzer G, Ranalter M, Wagner J, Glodny B, Hell T, Barnes T, Enk D. Individualised flow-controlled versus pressure-controlled ventilation in a porcine oleic acid-induced acute respiratory distress syndrome model. Eur J Anaesthesiol. 2023 Jul 1;40(7):511-520. doi: 10.1097/EJA.0000000000001807. Epub 2023 Feb 7. PMID 36749046
- [Background] Urner M, Juni P, Hansen B, Wettstein MS, Ferguson ND, Fan E. Time-varying intensity of mechanical ventilation and mortality in patients with acute respiratory failure: a registry-based, prospective cohort study. Lancet Respir Med. 2020 Sep;8(9):905-913. doi: 10.1016/S2213-2600(20)30325-8. Epub 2020 Jul 28. PMID 32735841
- [Background] Santer P, Wachtendorf LJ, Suleiman A, Houle TT, Fassbender P, Costa EL, Talmor D, Eikermann M, Baedorf-Kassis E, Schaefer MS. Mechanical Power during General Anesthesia and Postoperative Respiratory Failure: A Multicenter Retrospective Cohort Study. Anesthesiology. 2022 Jul 1;137(1):41-54. doi: 10.1097/ALN.0000000000004256. PMID 35475882
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367